CLINICAL TRIAL: NCT03405714
Title: A Multicenter, Open-Label Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of Intravenous Brivaracetam in Subjects >= 1 Month < 16 Years of Age With Epilepsy
Brief Title: A Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of Intravenous Brivaracetam in Subjects >= 1 Month to < 16 Years of Age With Epilepsy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCB Biopharma S.P.R.L. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EP0065; 2016-002452-25 (EudraCT Number)
Expanded Access: NCT03532516 (Available)
Record Dates: First submitted 2018-01-12; First posted 2018-01-23 (Actual); Results first posted 2021-11-26 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2021-12

CONDITIONS: Epilepsy
Keywords: Epilepsy; Brivaracetam; Briviact; Open-label; pediatric; intravenous
MeSH Terms: conditions — Epilepsy | interventions — brivaracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Brivaracetam (Experimental): Brivaracetam will be administered to various age-based cohorts. Cohort 1: Subjects >=12 to <16 years; Cohort 2: Subjects >=6 to <12 years; Cohort 3: Subjects >=2 to <6 years; Cohort 4: Subjects 1 month to <2 years. Enrollment will be sequential by descending age beginning with Cohort 1. For each cohort, the first half will receive a 15-minute iv infusion. The Data Monitoring Committee (DMC) will then review safety and, as available, PK data to make the following recommendations: the progression of the current cohort (up to 2-minute iv bolus infusion) and progression to initiate enrollment in the preceding cohort.
  Interventions: Drug: Brivaracetam

INTERVENTIONS:
Drug: Brivaracetam — * Pharmaceutical form: Solution for iv injection
  * Route of administration: intravenous use
  * Concentration: 10 mg/ml
  Other Names: Briviact

SUMMARY:
The purpose of the study is to evaluate the pharmacokinetics (PK), safety, and tolerability of brivaracetam (BRV) administered intravenously (iv) in subjects >= 1 month to < 16 years of age with epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female from >= 1 month to < 16 years of age. For subjects who are < 1 year from birth and who were preterm infants, the corrected gestational age should be used for this entry requirement
* Weight >= 3 kg (6.6 lbs)
* Diagnosis of epilepsy
* Acceptable candidate for venipuncture and intravenous (iv) infusion
* Treatment with >=1 anti epileptic drug (AED; including BRV) without a change of dose regimen for at least 7 days prior to Screening
* No treatment with vagus nerve stimulation (VNS), OR the subject is being treated with VNS and the settings have been constant for >=7 days prior to Screening
* For female subjects: not of childbearing potential, OR of childbearing potential and not sexually active/negative pregnancy test, OR of childbearing potential and sexually active/negative pregnancy test/uses medically acceptable contraceptive methods

Exclusion Criteria:

* Subject has previously received iv Brivaracetam (BRV) in this study
* Subject is being treated with BRV at a dose >5mg/kg/day (rounded) or >200mg/day for subjects with body weights >40kg
* Subject requires or is likely to require a change in concomitant antiepileptic drug(s) (AED[s]), dose of concomitant AED(s), or formulation of AED(s) during the 7 days prior to the intravenous (iv) pharmacokinetic (PK) Period
* Subject is likely, in the opinion of the Investigator, to require rescue medication during the Initiating Oral BRV (IOB) Treatment or iv PK Periods
* Subject has experienced generalized convulsive status epilepticus in the 28 days prior to Screening or during the Screening Period

Ages: 1 Month to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-11-04 (Actual); Study Completion 2020-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273 (UCB)
Locations (17):
- United States (2):
  - Ep0065 252, The Bronx, New York
  - Ep0065 237, Durham, North Carolina
- Czechia (2):
  - Ep0065 502, Hradec Králové
  - Ep0065 240, Prague
- Germany (2):
  - Ep0065 242, Berlin
  - Ep0065 254, Bielefeld
- Hungary (5):
  - Ep0065 210, Budapest
  - Ep0065 224, Budapest
  - Ep0065 247, Budapest
  - Ep0065 222, Debrecen
  - Ep0065 232, Miskolc
- Italy (4):
  - Ep0065 264, Milan
  - Ep0065 238, Pavia
  - Ep0065 239, Pavia
  - Ep0065 230, Roma
- Ep0065 223, Aguas Calientes, Mexico
- Ep0065 248, Seville, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Farkas MK, Kang H, Fogarasi A, Bozorg A, James GD, Krauwinkel W, Morita D, Will E, Elshoff JP. Pharmacokinetics, safety, and tolerability of intravenous brivaracetam in pediatric patients with epilepsy: An open-label trial. Epilepsia. 2022 Apr;63(4):855-864. doi: 10.1111/epi.17187. Epub 2022 Feb 23. PMID 35196395
- See also: Product Information — https://www.briviact.com/briviact-PI.pdf?v=1479491757
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll participants in June 2018 and concluded in November 2020.
Pre-assignment Details: Participant Flow refers to the Safety Set-Intravenous (SS-iv).
Groups:
- Age Cohort: >=12 to <16 Years: Screening Period (1-10 days): Participants receiving open-label BRV (OLB) or prescribed oral BRV (RxB) continued to receive oral BRV. IOB Treatment Period (2-10 days): Participants who initiated Oral BRV (IOB) continued with oral BRV 2 milligram/kilogram/day (mg/kg/day). IV PK (Intravenous Pharmacokinetic) Period (1-6 days): During iv PK Period, iv BRV was administered every 12 hours. For OLB, RxB, and IOB participants, first iv Brivaracetam (BRV) dose was equivalent to final dose of oral BRV and for Initiating iv BRV (IIB) participants, first iv BRV dose was 1mg/kg. For each cohort, the first half received 15-minute infusion, the remaining half as a bolus (up to 2-minute infusion). Down-Titration Period: Participants who discontinued treatment, had their BRV dose reduced every week for a maximum of 4 weeks down to a dose of 1mg/kg/day.
- Age Cohort: >=6 to <12 Years; Age Cohort: >=2 to <6 Years; Age Cohort: >=1 Month to <2 Years: Screening Period (1-10 days): Participants receiving OLB or RxB continued to receive oral BRV. IOB Treatment Period (2-10 days): IOB Participants continued with oral BRV 2mg/kg/day. IV PK Period (1-6 days): During iv PK Period, iv BRV was administered every 12 hours. For OLB, RxB, and IOB participants, first iv BRV dose was equivalent to final dose of oral BRV and for IIB participants, first iv BRV dose was 1mg/kg. For each cohort, the first half received the 15-minute infusion, the remaining half as a bolus (up to 2-minute infusion). Down-Titration Period: Participants who discontinued treatment, had their BRV dose reduced every week for a maximum of 4 weeks down to a dose of 1mg/kg/day.
Period: Overall Study
Arm/Group | Age Cohort: >=12 to <16 Years | Age Cohort: >=6 to <12 Years | Age Cohort: >=2 to <6 Years | Age Cohort: >=1 Month to <2 Years
Started | 12 | 12 | 13 | 13
Completed | 12 | 12 | 13 | 13
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to SS-iv, which included study participants who received at least 1 dose of iv BRV.
Arm/Group | Age Cohort: >=12 to <16 Years | Age Cohort: >=6 to <12 Years | Age Cohort: >=2 to <6 Years | Age Cohort: >=1 Month to <2 Years | Total Title
Number analyzed (Participants) | 12 | 12 | 13 | 13 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 12 | 12 | 13 | 13 | 50
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.08 (1.16) | 8.33 (1.61) | 3.85 (0.99) | 0.95 (0.59) | 6.39 (4.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 5 | 5 | 24
  Male | 6 | 4 | 8 | 8 | 26
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian/Alaskan Native | 0 | 0 | 0 | 2 | 2
  Black | 1 | 0 | 0 | 0 | 1
  White | 11 | 12 | 13 | 11 | 47

OUTCOME MEASURES:

1. Primary Outcome: Plasma Concentration of Brivaracetam (BRV) at Predose (<=1 Hour), Visit 3
Description: Blood samples were taken at indicated time points to determine brivaracetam (BRV) plasma concentration before, during, and after iv BRV administration.
Time Frame: Blood samples were collected at <= 1 hour pre-initiation of intravenous (iv) BRV infusion at Visit 3 (Day 1 of IV PK period)
Population: The PK-PPS included all study participants in the SS-iv having provided at least 1 measurable postdose plasma sample (with recorded sampling time) during the iv PK Period with documented iv BRV infusion times and without IPDs impacting the interpretability of the PK analyses. Here, N (number of participants analyzed) were included who were evaluable for the assessment.
Measure: Geometric Mean (95% Confidence Interval); unit: nanograms per milliliter (ng/mL)
Groups:
- Age Cohort: >=12 to <16 Years (PK-PPS): Participants received iv administration of BRV every 12 hours during the IV PK Period (1-6days). For OLB, RxB, and IOB participants, first iv BRV dose was equivalent to final dose of oral BRV and for IIB participants, first iv BRV dose was 1mg/kg. For each cohort, the first half received the 15-minute infusion, the remaining as a bolus (up to 2-minute infusion). Participants formed the Pharmacokinetic Per-protocol Set (PK-PPS).
- Age Cohort: >=6 to <12 Years (PK-PPS); Age Cohort: >=2 to <6 Years (PK-PPS); Age Cohort : >=1 Month to <2 Years (PK-PPS): Participants received iv administration of BRV every 12 hours during the IV PK Period (1-6days). For OLB, RxB, and IOB participants, first iv BRV dose was equivalent to final dose of oral BRV and for IIB participants, first iv BRV dose was 1mg/kg. For each cohort, the first half received the 15-minute infusion, the remaining as a bolus (up to 2-minute infusion). Participants formed the PK-PPS.
Arm/Group | Age Cohort: >=12 to <16 Years (PK-PPS) | Age Cohort: >=6 to <12 Years (PK-PPS) | Age Cohort: >=2 to <6 Years (PK-PPS) | Age Cohort : >=1 Month to <2 Years (PK-PPS)
Number analyzed (Participants) | 12 | 10 | 10 | 9
nanograms per milliliter (ng/mL) | 149.0 [27.6 to 805.1] | NA [NA to NA] — Geometric mean and 95% CI were only calculated if at least two-thirds of the data were greater than the lower Limit of quantification (LOQ). | NA [NA to NA] — Geometric mean and 95% CI were only calculated if at least two-thirds of the data were greater than the lower Limit of quantification (LOQ). | 310.6 [92.5 to 1042.7]

2. Primary Outcome: Plasma Concentration of Brivaracetam (BRV) at Postdose 15 Minutes, Visit 3
Description: as for outcome 1
Time Frame: Blood samples were collected at 15 minutes post-initiation of iv BRV infusion at Visit 3 (Day 1 of IV PK period)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Age Cohort: >=12 to <16 Years (PK-PPS) | Age Cohort: >=6 to <12 Years (PK-PPS) | Age Cohort: >=2 to <6 Years (PK-PPS) | Age Cohort : >=1 Month to <2 Years (PK-PPS)
Number analyzed (Participants) | 12 | 10 | 8 | 10
ng/mL | 1844.6 [1110.4 to 3064.3] | 2058.8 [1726.4 to 2455.2] | 1774.9 [1087.4 to 2897.1] | 1566.6 [973.1 to 2522.2]

3. Primary Outcome: Plasma Concentration of Brivaracetam (BRV) at Postdose 3 Hours, Visit 3
Description: as for outcome 1
Time Frame: Blood samples were collected at 3 hours post-initiation of iv BRV infusion at Visit 3 (Day 1 of IV PK period)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Age Cohort: >=12 to <16 Years (PK-PPS) | Age Cohort: >=6 to <12 Years (PK-PPS) | Age Cohort: >=2 to <6 Years (PK-PPS) | Age Cohort : >=1 Month to <2 Years (PK-PPS)
Number analyzed (Participants) | 12 | 10 | 11 | 9
ng/mL | 1260.6 [962.6 to 1650.8] | 1189.5 [1005.5 to 1407.1] | 1225.3 [676.8 to 2218.6] | 1341.7 [657.9 to 2735.9]

4. Primary Outcome: Plasma Concentration of Brivaracetam (BRV) at Predose (<=1 Hour), Visit 4
Description: as for outcome 1
Time Frame: Blood samples were collected at <= 1 hour pre-initiation of intravenous (iv) BRV infusion at Visit 4 (Day 2 of IV PK period)
Population: The PK-PPS included all study participants in the SS-iv having provided at least 1 measurable postdose plasma sample (with recorded sampling time) during the iv PK Period with documented iv BRV infusion times and without IPDs impacting the interpretability of the PK analyses. Here, N (number of participants analyzed) were included who were evaluable for the assessment. PK samples were not collected at Visit 4 in >=12 to <16 years, >=2 to <6 years, and >=1 to <2 years patients.
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Age Cohort: >=12 to <16 Years (PK-PPS) | Age Cohort: >=6 to <12 Years (PK-PPS) | Age Cohort: >=2 to <6 Years (PK-PPS) | Age Cohort : >=1 Month to <2 Years (PK-PPS)
Number analyzed (Participants) | 0 | 3 | 0 | 0
ng/mL |  | 290.5 [101.2 to 834.0] |  |

5. Primary Outcome: Plasma Concentration of Brivaracetam (BRV) at Postdose 15 Minutes, Visit 4
Description: as for outcome 1
Time Frame: Blood samples were collected at 15 minutes post-initiation of iv BRV infusion at Visit 4 (Day 2 of IV PK period)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Age Cohort: >=12 to <16 Years (PK-PPS) | Age Cohort: >=6 to <12 Years (PK-PPS) | Age Cohort: >=2 to <6 Years (PK-PPS) | Age Cohort : >=1 Month to <2 Years (PK-PPS)
Number analyzed (Participants) | 0 | 3 | 0 | 0
ng/mL |  | 2084.3 [681.2 to 6377.0] |  |

6. Primary Outcome: Plasma Concentration of Brivaracetam (BRV) at Postdose 3 Hours, Visit 4
Description: as for outcome 1
Time Frame: Blood samples were collected at 3 hours post-initiation of iv BRV infusion at Visit 4 (Day 2 of IV PK period)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Age Cohort: >=12 to <16 Years (PK-PPS) | Age Cohort: >=6 to <12 Years (PK-PPS) | Age Cohort: >=2 to <6 Years (PK-PPS) | Age Cohort : >=1 Month to <2 Years (PK-PPS)
Number analyzed (Participants) | 0 | 3 | 0 | 0
ng/mL |  | 1149.8 [613.1 to 2156.4] |  |

7. Primary Outcome: Plasma Concentration of Brivaracetam (BRV) at Predose (<=1 Hour), Visit 5
Description: as for outcome 1
Time Frame: Blood samples were collected at <= 1 hour pre-initiation of intravenous (iv) BRV infusion at Visit 5 (Day 2 of IV PK period)
Population: The PK-PPS included all study participants in the SS-iv having provided at least 1 measurable postdose plasma sample (with recorded sampling time) during the iv PK Period with documented iv BRV infusion times and without IPDs impacting the interpretability of the PK analyses. Here, N (number of participants analyzed) were included who were evaluable for the assessment. PK samples were not collected at Visit 5 in >=12 to <16 years patients.
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Age Cohort: >=12 to <16 Years (PK-PPS) | Age Cohort: >=6 to <12 Years (PK-PPS) | Age Cohort: >=2 to <6 Years (PK-PPS) | Age Cohort : >=1 Month to <2 Years (PK-PPS)
Number analyzed (Participants) | 0 | 1 | 2 | 3
ng/mL |  | 466.0 [NA to NA] — 'NA' signifies that 95% CI could not be calculated for a single participant. | 204.5 [0.1 to 383063.7] | 482.9 [4.8 to 48506.1]

8. Primary Outcome: Plasma Concentration of Brivaracetam (BRV) at Postdose 15 Minutes, Visit 5
Description: as for outcome 1
Time Frame: Blood samples were collected at 15 minutes post-initiation of iv BRV infusion at Visit 5 (Day 2 of IV PK period)
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Age Cohort: >=12 to <16 Years (PK-PPS) | Age Cohort: >=6 to <12 Years (PK-PPS) | Age Cohort: >=2 to <6 Years (PK-PPS) | Age Cohort : >=1 Month to <2 Years (PK-PPS)
Number analyzed (Participants) | 0 | 1 | 3 | 3
ng/mL |  | 2890.0 [NA to NA] — 'NA' signifies that 95% CI could not be calculated for a single participant. | 1948.8 [690.8 to 5497.7] | 2072.4 [743.2 to 5778.8]

9. Primary Outcome: Plasma Concentration of Brivaracetam (BRV) at Postdose 3 Hours, Visit 5
Description: as for outcome 1
Time Frame: Blood samples were collected at 3 hours post-initiation of iv BRV infusion at Visit 5 (Day 2 of IV PK period)
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Age Cohort: >=12 to <16 Years (PK-PPS) | Age Cohort: >=6 to <12 Years (PK-PPS) | Age Cohort: >=2 to <6 Years (PK-PPS) | Age Cohort : >=1 Month to <2 Years (PK-PPS)
Number analyzed (Participants) | 0 | 1 | 2 | 3
ng/mL |  | 1820 [NA to NA] — 'NA' signifies that 95% CI could not be calculated for a single participant. | 1203.5 [147.1 to 9847.1] | 727.4 [144.9 to 3652.9]

10. Primary Outcome: Plasma Concentration of Brivaracetam (BRV) at Predose (<=1 Hour), Visit 3 by Infusion Duration - 15 Minutes
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Groups:
- 15-minute Infusion (PK-PPS): Participants received iv administration of BRV every 12 hours during the IV PK Period (1-6 days). For OLB, RxB, and IOB participants, first iv BRV dose was equivalent to final dose of oral BRV and for IIB participants, first iv BRV dose was 1mg/kg. For each cohort, the first half received the 15-minute infusion. Participants formed the PK-PPS.
Arm/Group | 15-minute Infusion (PK-PPS)
Number analyzed (Participants) | 19
ng/mL | NA [NA to NA] — Geometric mean and 95% CI were only calculated if at least two-thirds of the data were greater than the lower Limit of quantification (LOQ).

11. Primary Outcome: Plasma Concentration of Brivaracetam (BRV) at Postdose 15 Minutes, Visit 3 by Infusion Duration- 15 Minutes
Description: as for outcome 1
Time Frame: Blood samples were collected at 15 minutes post-initiation of iv BRV infusion at Visit 3 (Day 1 of IV PK period)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | 15-minute Infusion (PK-PPS)
Number analyzed (Participants) | 21
ng/mL | 1903.0 [1474.9 to 2455.4]

12. Primary Outcome: Plasma Concentration of Brivaracetam (BRV) at Postdose 3 Hours, Visit 3 by Infusion Duration- 15 Minutes
Description: as for outcome 1
Time Frame: Blood samples were collected at 3 hours post-initiation of iv BRV infusion at Visit 3 (Day 1 of IV PK period)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | 15-minute Infusion (PK-PPS)
Number analyzed (Participants) | 21
ng/mL | 1130.3 [882.1 to 1448.3]

13. Primary Outcome: Plasma Concentration of Brivaracetam (BRV) at Predose (<=1 Hour), Visit 4 by Infusion Duration- 15 Minutes
Description: as for outcome 1
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | 15-minute Infusion (PK-PPS)
Number analyzed (Participants) | 3
ng/mL | 290.5 [101.2 to 834.0]

14. Primary Outcome: Plasma Concentration of Brivaracetam (BRV) at Postdose 15 Minutes, Visit 4 by Infusion Duration- 15 Minutes
Description: as for outcome 1
Time Frame: Blood samples were collected at 15 minutes post-initiation of iv BRV infusion at Visit 4 (Day 2 of IV PK period)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | 15-minute Infusion (PK-PPS)
Number analyzed (Participants) | 3
ng/mL | 2084.3 [681.2 to 6377.0]

15. Primary Outcome: Plasma Concentration of Brivaracetam (BRV) at Postdose 3 Hours, Visit 4 by Infusion Duration- 15 Minutes
Description: as for outcome 1
Time Frame: Blood samples were collected at 3 hours post-initiation of iv BRV infusion at Visit 4 (Day 2 of IV PK period)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | 15-minute Infusion (PK-PPS)
Number analyzed (Participants) | 3
ng/mL | 1149.8 [613.1 to 2156.4]

16. Primary Outcome: Plasma Concentration of Brivaracetam (BRV) at Predose (<=1 Hour), Visit 5 by Infusion Duration- 15 Minutes
Description: as for outcome 1
Time Frame: as for outcome 7
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | 15-minute Infusion (PK-PPS)
Number analyzed (Participants) | 3
ng/mL | 776.0 [51.9 to 11611.3]

17. Primary Outcome: Plasma Concentration of Brivaracetam (BRV) at Postdose 15 Minutes, Visit 5 by Infusion Duration- 15 Minutes
Description: as for outcome 1
Time Frame: Blood samples were collected at 15 minutes post-initiation of iv BRV infusion at Visit 5 (Day 2 of IV PK period)
Population: The PK-PPS included all study participants in the SS-iv having provided at least 1 measurable postdose plasma sample (with recorded sampling time) during the iv PK Period with documented iv BRV infusion times and without IPDs impacting the interpretability of the PK analyses.
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | 15-minute Infusion (PK-PPS)
Number analyzed (Participants) | 4
ng/mL | 2697.8 [1911.1 to 3808.3]

18. Primary Outcome: Plasma Concentration of Brivaracetam (BRV) at Postdose 3 Hours, Visit 5 by Infusion Duration- 15 Minutes
Description: as for outcome 1
Time Frame: Blood samples were collected at 3 hours post-initiation of iv BRV infusion at Visit 5 (Day 2 of IV PK period)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | 15-minute Infusion (PK-PPS)
Number analyzed (Participants) | 4
ng/mL | 1030.0 [376.1 to 2820.9]

19. Primary Outcome: Plasma Concentration of Brivaracetam (BRV) at Predose (<=1 Hour), Visit 3 by Infusion Duration- Bolus
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 17
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Groups:
- Bolus (PK-PPS): Participants received iv administration of BRV every 12 hours during the IV PK Period (1-6days). For OLB, RxB, and IOB participants, first iv BRV dose was equivalent to final dose of oral BRV and for IIB participants, first iv BRV dose was 1mg/kg. For each cohort the second half received the bolus (up to 2-minute infusion). Participants formed PK-PPS.
Arm/Group | Bolus (PK-PPS)
Number analyzed (Participants) | 22
ng/mL | 120.5 [44.7 to 325.2]

20. Primary Outcome: Plasma Concentration of Brivaracetam (BRV) at Postdose 15 Minutes, Visit 3 by Infusion Duration- Bolus
Description: as for outcome 1
Time Frame: Blood samples were collected at 15 minutes post-initiation of iv BRV infusion at Visit 3 (Day 1 of IV PK period)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Bolus (PK-PPS)
Number analyzed (Participants) | 19
ng/mL | 1704.8 [1237.5 to 2348.4]

21. Primary Outcome: Plasma Concentration of Brivaracetam (BRV) at Postdose 3 Hours, Visit 3 by Infusion Duration- Bolus
Description: as for outcome 1
Time Frame: Blood samples were collected at 3 hours post-initiation of iv BRV infusion at Visit 3 (Day 1 of IV PK period)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Bolus (PK-PPS)
Number analyzed (Participants) | 21
ng/mL | 1383.9 [989.3 to 1935.8]

22. Primary Outcome: Plasma Concentration of Brivaracetam (BRV) at Predose (<=1 Hour), Visit 4 by Infusion Duration- Bolus
Description: as for outcome 1
Time Frame: At <= 1 hour pre-initiation of intravenous (iv) BRV infusion at Visit 4 (Day 2 of IV PK period)
Population: The PK-PPS included all study participants in the SS-iv having provided at least 1 measurable postdose plasma sample (with recorded sampling time) during the iv PK Period with documented iv BRV infusion times and without IPDs impacting the interpretability of the PK analyses. PK samples were not collected at Visit 4 in bolus patients.
Arm/Group | Bolus (PK-PPS)
Number analyzed (Participants) | 0

23. Primary Outcome: Plasma Concentration of Brivaracetam (BRV) at Postdose 15 Minutes, Visit 4 by Infusion Duration- Bolus
Description: as for outcome 1
Time Frame: At 15 minutes post-initiation of iv BRV infusion at Visit 4 (Day 2 of IV PK period)
Population: as for outcome 22
Arm/Group | Bolus (PK-PPS)
Number analyzed (Participants) | 0

24. Primary Outcome: Plasma Concentration of Brivaracetam (BRV) at Postdose 3 Hours, Visit 4 by Infusion Duration- Bolus
Description: as for outcome 1
Time Frame: At 3 hours post-initiation of iv BRV infusion at Visit 4 (Day 2 of IV PK period)
Population: as for outcome 22
Arm/Group | Bolus (PK-PPS)
Number analyzed (Participants) | 0

25. Primary Outcome: Plasma Concentration of Brivaracetam (BRV) at Predose (<=1 Hour), Visit 5 by Infusion Duration- Bolus
Description: as for outcome 1
Time Frame: as for outcome 7
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Bolus (PK-PPS)
Number analyzed (Participants) | 3
ng/mL | 167.5 [9.6 to 2932.2]

26. Primary Outcome: Plasma Concentration of Brivaracetam (BRV) at Postdose 15 Minutes, Visit 5 by Infusion Duration- Bolus
Description: as for outcome 1
Time Frame: Blood samples were collected at 15 minutes post-initiation of iv BRV infusion at Visit 5 (Day 2 of IV PK period)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Bolus (PK-PPS)
Number analyzed (Participants) | 3
ng/mL | 1531.8 [837.3 to 2802.2]

27. Primary Outcome: Plasma Concentration of Brivaracetam (BRV) at Postdose 3 Hours, Visit 5 by Infusion Duration- Bolus
Description: as for outcome 1
Time Frame: Blood samples were collected at 3 hours post-initiation of iv BRV infusion at Visit 5 (Day 2 of IV PK period)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Bolus (PK-PPS)
Number analyzed (Participants) | 2
ng/mL | 949.5 [2.8 to 316987.2]

28. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: An adverse event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product that does not necessarily have a causal relationship with this treatment.
Time Frame: From Screening until last visit (up to Day 68)
Population: The SS-iv included study participants who received at least 1 dose of iv BRV.
Measure: Count of Participants; unit: Participants
Groups:
- Age Cohort: >=12 to <16 Years (SS-iv): Screening Period (1-10 days): Participants receiving OLB or RxB continued to receive oral BRV. IOB Treatment Period (2-10 days): IOB Participants continued with oral BRV 2mg/kg/day. IV PK Period (1-6 days): During iv PK Period, iv BRV was administered every 12 hours. For OLB, RxB, and IOB participants, first iv BRV dose was equivalent to final dose of oral BRV and for IIB participants, first iv BRV dose was 1mg/kg. For each cohort, the first half received the 15-minute infusion, the remaining half as a bolus (up to 2-minute infusion). Down-Titration Period: Participants who discontinued treatment, had their BRV dose reduced every week for a maximum of 4 weeks down to a dose of 1mg/kg/day. Participants formed the Safety Set-Intravenous (SS-iv).
- Age Cohort: >=6 to <12 Years (SS-iv); Age Cohort: >=1 Month to <2 Years (SS-iv): Screening Period (1-10 days): Participants receiving OLB or RxB continued to receive oral BRV. IOB Treatment Period (2-10 days): IOB Participants continued with oral BRV 2mg/kg/day. IV PK Period (1-6 days): During iv PK Period, iv BRV was administered every 12 hours. For OLB, RxB, and IOB participants, first iv BRV dose was equivalent to final dose of oral BRV and for IIB participants, first iv BRV dose was 1mg/kg. For each cohort, the first half received the 15-minute infusion, the remaining half as a bolus (up to 2-minute infusion). Down-Titration Period: Participants who discontinued treatment, had their BRV dose reduced every week for a maximum of 4 weeks down to a dose of 1mg/kg/day. Participants formed the SS-iv.
- Age Cohort: >=2 to <6 Years (SS-iv): Screening Period (1-10 days): Participants receiving OLB or RxB continued to receive oral BRV. IOB Treatment Period (2-10 days): IOB Participants continued with oral BRV 2mg/kg/day. IV PK Period (1-6 days): During iv PK Period, iv BRV was administered every 12 hours. For OLB, RxB, and IOB participants, first iv BRV dose was equivalent to final dose of oral BRV and for IIB participants, first iv BRV dose was 1mg/kg. For each cohort, the first half received the 15-minute infusion, the remaining half as a bolus (up to 2-minute infusion). Down-Titration Period: Participants who discontinued treatment, had their BRV dose reduced every week for a maximum of 4 weeks down to a dose of 1mg/kg/day. Participants formed the Safety SS-iv.
Arm/Group | Age Cohort: >=12 to <16 Years (SS-iv) | Age Cohort: >=6 to <12 Years (SS-iv) | Age Cohort: >=2 to <6 Years (SS-iv) | Age Cohort: >=1 Month to <2 Years (SS-iv)
Number analyzed (Participants) | 12 | 12 | 13 | 13
Participants | 3 | 4 | 7 | 2

29. Primary Outcome: Number of Participant Withdrawals Due to Adverse Events
Description: as for outcome 28
Time Frame: From Screening until last visit (up to Day 68)
Population: The SS-iv included study participants who received at least 1 dose of iv BRV.
Measure: Count of Participants; unit: Participants
Arm/Group | Age Cohort: >=12 to <16 Years (SS-iv) | Age Cohort: >=6 to <12 Years (SS-iv) | Age Cohort: >=2 to <6 Years (SS-iv) | Age Cohort: >=1 Month to <2 Years (SS-iv)
Number analyzed (Participants) | 12 | 12 | 13 | 13
Participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From Screening until last visit (up to Day 68)
Arm/Group | Age Cohort: >=12 to <16 Years (SS-iv) | Age Cohort: >=6 to <12 Years (SS-iv) | Age Cohort: >=2 to <6 Years (SS-iv) | Age Cohort: >=1 Month to <2 Years (SS-iv)
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/13 | 1/13
Other Adverse Events (participants affected / at risk) | 3/12 | 4/12 | 7/13 | 2/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Age Cohort: >=12 to <16 Years (SS-iv) (N=12) | Age Cohort: >=6 to <12 Years (SS-iv) (N=12) | Age Cohort: >=2 to <6 Years (SS-iv) (N=13) | Age Cohort: >=1 Month to <2 Years (SS-iv) (N=13)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Age Cohort: >=12 to <16 Years (SS-iv) (N=12) | Age Cohort: >=6 to <12 Years (SS-iv) (N=12) | Age Cohort: >=2 to <6 Years (SS-iv) (N=13) | Age Cohort: >=1 Month to <2 Years (SS-iv) (N=13)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Vessel puncture site haemorrhage (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Aggression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-06-19): https://cdn.clinicaltrials.gov/large-docs/14/NCT03405714/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-25): https://cdn.clinicaltrials.gov/large-docs/14/NCT03405714/SAP_001.pdf